CLINICAL TRIAL: NCT07275034
Title: A Virtual Reality-Based Horticultural Planting Program for Elderly With Subthreshold Depression：A Randomized Controlled Pilot Study
Brief Title: A Virtual Reality-Based Horticultural Planting Program for Elderly With Subthreshold Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Zhu Ziping, Study Director, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: K2025-06-025
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Subthreshold Depression
Keywords: older adults; Subthreshold Depression; virutal reality; Gardening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Intervention (Experimental): This group utilized a virtual reality intervention system based on horticultural planting, designed and developed by the research team.
  Interventions: Other: Virtual Reality Garden System
- Routine Care (Experimental): This arm of seniors maintains their daily routines and participates regularly in the nursing home's daily activities.
  Interventions: Other: Routine Care

INTERVENTIONS:
Other: Virtual Reality Garden System — The system comprised six tasks. Task One was an individual task involving planting tomatoes by completing eight subtasks (tilling, sowing, fertilizing, watering, secondary fertilization, secondary watering, pest control, harvesting) in a virtual garden. Tasks Two through Five were two-player online cooperative tasks. Task 2 involves corn cultivation, with one participant planting while the other observes; Task 3 requires two participants to simultaneously plant strawberries in parallel within the virtual garden; Task 4 involves collaborative sunflower planting between two participants; Task 5 has experienced elderly participants assisting less experienced individuals in completing planting tasks; Task 6 enables three participants to share the joy of planting together in the virtual garden.
  Arms: Virtual Reality Intervention
Other: Routine Care — This arm of seniors maintains their daily routines and participates regularly in the nursing home's daily activities.
  Arms: Routine Care

SUMMARY:
Subthreshold depression represents a state of psychological sub-health between normal individuals and clinical depression. It constitutes a high-risk stage for developing clinical depression and a critical phase for alleviating depressive symptoms. However, current research predominantly focuses on treating depression in the elderly, with insufficient attention to interventions for high-risk populations or limited to cross-sectional investigations of subthreshold depression risk factors. Therefore, prioritizing subthreshold depression in the elderly and implementing early interventions is essential. A 2024 article in The Lancet suggests that subthreshold depression treatment should prioritize psychotherapy and lifestyle adjustments over medication. Horticultural therapy, an interdisciplinary approach integrating horticulture, medicine, and psychology, demonstrates unique advantages over traditional medical treatments. In practical application, however, limited resources may hinder adequate support for horticultural activities, compromising activity quality, reducing therapeutic efficacy, and restricting the widespread adoption of horticultural therapy. Integrating VR technology with horticultural therapy can provide patients with more comprehensive, personalized, and effective mental health treatment plans, empowering them toward healthier, more positive lives. Therefore, the research team designed a VR horticultural intervention system for elderly individuals with subthreshold depression based on the Social Participation Competence Framework.

DETAILED DESCRIPTION:
Subthreshold depression (SD) represents a state of psychological sub-health between normal individuals and clinical depression. It constitutes a high-risk stage for developing major depressive disorder and a critical window for alleviating depressive symptoms. An editorial published in JAMA emphasized that research on subthreshold depression holds significant implications for exploring the prevention and treatment of depression. Therefore, prioritizing subthreshold depression in older adults and implementing early interventions is essential. Multiple studies indicate that social engagement, as one of the modifiable factors for depression in older adults, can actively delay the onset and progression of geriatric depression. Social engagement encompasses multidimensional activities through which older adults exchange material and emotional resources and gain social recognition. These include participation in activities, fulfillment of social roles, interpersonal interactions, utilization of social resources, and the restoration of personal value. Factors such as retirement, illness, or physical decline often lead to a narrowing of older adults' existing social networks and weakened social connections. This results in reduced scope and frequency of social engagement, potentially triggering or exacerbating depressive disorders. Conversely, depressive disorders themselves, through core symptoms like low mood and diminished interest, further undermine older adults' willingness and ability to maintain relationships and actively participate in activities, creating a vicious cycle. A 2024 study published in The Lancet indicates that older adults with high levels of social engagement exhibit significantly lower depression risk compared to those with low engagement. Similarly, a 2023 Nature Aging study suggests that social participation may reduce depression by alleviating stress, inflammation, and cerebrovascular damage, thereby preserving brain health, building cognitive reserve, and mitigating depressive disorders.

Virtual Reality (VR) technology, as a novel intervention method, possesses three key characteristics: immersion, interactivity, and simulation. By replicating real-world settings such as home and community environments, it enriches the training experience for elderly individuals with depression, helping them adapt to diverse social contexts and enhancing intervention outcomes. Horticultural therapy, an interdisciplinary approach integrating horticulture, medicine, and psychology, offers relatively low treatment costs with minimal side effects. It plays a positive role in promoting physical recovery, improving emotional well-being, and enhancing social skills. Increasingly, research teams are exploring VR-generated virtual horticultural environments and horticultural activity interventions. VR technology addresses multiple limitations of traditional horticultural therapy. VR-based gardening activities overcome temporal and spatial constraints, reduce the costs and risks associated with physical gardening, and provide richer, more personalized socialized horticultural settings and activities that cater to diverse patient needs. Therefore, integrating VR technology with horticultural therapy offers patients a more comprehensive, personalized, and effective mental health treatment plan, empowering them to lead healthier, more positive lives.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Meets subthreshold depression diagnostic criteria: CES-D score ≥ 16 on the Center for Epidemiological Survey, Depression Scale (CES-D) used in epidemiological surveys (this criterion is widely adopted in comparable studies)
* No communication barriers in vision, hearing, or speech
* Informed consent

Exclusion Criteria:

* Insulin dependent diabetes
* Thyroid disease
* Recent exposure to a major traumatic stress event, with no risk of suicide
* Currently participating in other similar studies
* Clinically diagnosed with mental disorders such as depression or schizophrenia
* Currently taking antidepressant medication
* Severe cognitive impairment
* Severe physical illness or organic disorder with impaired self-care abilities

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Subthreshold Depression | The intervention was conducted in November 2025, and the evaluation time was 0,4,9 weeks .
  The Center for Epidemiological Surveys Depression Scale (CES-D) was developed by Rirodiff at the National Institute of Mental Health in the United States. It is designed for screening depressive symptoms in older adults, comprising 20 items. Each question assesses one symptom, covering 20 distinct symptoms in total. The total score ranges from 0 to 60 points. A score ≤15 indicates no depressive symptoms, 16-19 suggests possible depressive symptoms, and ≥20 confirms depressive symptoms. The Cronbach's alpha coefficient for the Chinese population is 0.90. It is one of the most commonly used subthreshold depression epidemiological survey tools, with existing studies defining CES-D ≥16 as subthreshold depression.
  Translated with DeepL.com (free version)

SECONDARY OUTCOMES:
General cognitive function | The intervention was conducted in September 2025, and the evaluation time was 0,4,9 weeks separately.
  The Montreal Coanitive Asessment Scale,developed by Nasreddine in 2004 to assess participants'general cognitive function, covers eight areasof cognitive assessment, including visuospatial and executive function, naming, memory, attention, speech, abstraction, delayed recall, andorientation. The Changsha version of the Montreal Cognitive Assessment Scale was used in this study, and its Cronbach's a coeficient was 0.846,retest reliability was 0.974, and investigator reliability was 0.969. The score of the Montreal Cognitive Assessment Scale ranges from 0 to 30points. The higher the score,the better the cognitive function ofthe study subjects. The iliterate group s13, the primary school group s19 and thejunior high school and above group s24 can be judged as impaired cognitive function to correct the bias caused by education level.
Anxiety Condition | The intervention was conducted in November 2025, and the evaluation time was 0,4,9 weeks separately
  The self-rating anxiety scale (SAS) was designed and developed by Zung in the United States in 1971 to assess the severity of anxiety symptoms in individuals. It demonstrates good reliability and validity, with a split-half reliability coefficient of 0.696, test-retest reliability of 0.777, and internal consistency of 0.82. Additionally, it exhibits good construct validity . The scale comprises 20 items, with items 5, 9, 13, 17, and 19 scored in reverse. The scale employs a 1-4 rating scale (1 = never or rarely; 2 = a small portion of the time; 3 = a considerable portion of the time; 4 = most or all of the time). Individuals complete the scale based on their experiences during the past week. The total score is multiplied by 1.25, rounded to the nearest whole number to obtain a standardized score, which serves as the statistical indicator. A higher standardized score indicates more severe anxiety levels
Activities of Daily Living | The intervention was conducted in September 2025, and the evaluation time was 0,4,9 weeks separately.
  This study employs the Activities of Daily Living (ADL) scale developed by Lawton and Brody in 1969 to assess an individual's self-care abilities and functional status in daily life. The version selected for this study, adapted into Chinese by Zhang Mingyuan et al., comprises 20 items using a 4-point Likert scale. The total score ranges from 20 to 80 points, with higher scores indicating poorer ability to perform activities of daily living. The Cronbach's α coefficient for this scale is 0.92.
Social Support | The intervention was conducted in September 2025, and the evaluation time was 0,4,9 weeks separately.
  Social Support Rating Scale (SSRS) This study employed the SSRS developed by Xiao Shuiyuan in 1986 to assess patients' levels of social support. The scale comprises three dimensions: objective support (3 items), subjective support (4 items), and utilization of support (3 items), totaling 20 items. Items 1, 4, 5, 6, 8, 9, and 10 are single-choice questions. Options (1), (2), (3), (4) are scored as 1, 2, 3, and 4 points respectively. For items 2 and 3, the "No sources at all" option scores 0 points, while the "The following sources" option scores points corresponding to the number of sources selected. In item 7, options A, B, C, D, and E are scored from 1 to 4 points, ranging from 'None' to "Full support," respectively. The total score ranges from 12 to 66 points. Higher scores indicate greater levels of social support for the patient. The Cronbach's α coefficient for this scale ranges from 0.89 to 0.94.
Sleep Quality | The intervention was conducted in September 2025, and the evaluation time was 0,4,9 weeks separately.
  This study employed the Pittsburgh Sleep Quality Index (PSQI) developed by Buysse et al. in 1989 to assess patients' sleep quality over the preceding month. The 19-item questionnaire comprises seven components: subjective sleep quality, sleep onset latency, sleep duration, sleep efficiency, sleep disturbances, hypnotic medication use, and daytime functioning. The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality. The Cronbach's alpha coefficient for this scale is 0.85.
System Usability | The intervention will be implemented in November 2025, with the evaluation conducted after the 9-week intervention period concludes.
  System Usability Scale (SUS) Developed by Brooke et al., the scale used in this study is the Chinese version of the System Usability Scale translated and revised by Chinese scholars including Li Yongfeng. This scale is unidimensional and consists of 10 items. It employs a 5-point Likert scale, with scores ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). Positive items (Items 1, 3, 5, 7, 9) are scored positively: Actual item score = Item rating - 1. Negative items (Items 2, 4, 6, 8, 10) are scored negatively: Actual item score = 5 - Item rating. If an item is left blank, it is assigned a score of 3. The total scale score = sum of all item scores × 2.5. The scale has a maximum score of 100 points, with scores >60 considered usable, 70 considered good, ≥80 considered excellent, and ≥90 considered outstanding. The Cronbach's alpha coefficient for this scale is 0.91.
Simulator Sickness | The intervention will be implemented in November 2025, with the evaluation conducted after the 9-week intervention period concludes.
  The Simulator Sickness Questionnaire(SSQ) developed by Kennedy et al. in 1993, is a widely used tool for assessing the subjective severity of simulator sickness symptoms. The SSQ consists of pre- and post-experiment sections. The pre-experiment section employs the Pensacola Motion Sickness Questionnaire (MSQ) to gather information about participants' current physical condition and prior simulator experience. The post-experiment section measures symptom severity on a four-point scale (0-3) for each symptom. SSQ items can be grouped into three factors: nausea (e.g., sweating, difficulty concentrating, gastric awareness), eye movement disturbances (e.g., headache, eye fatigue, blurred vision), and disorientation (e.g., head fullness, dizziness with eyes open/closed, vertigo). The SSQ can be scored in two ways: (1) Calculate the score for each factor by summing the scores of all relevant items (each factor includes 7 items), with a score range of 0-179.5
Immersion Presence | The intervention will be implemented in November 2025, with the evaluation conducted after the 9-week intervention period concludes.
  The Immersion Presence Questionnaire (IPQ) was employed to evaluate users' sense of immersion in the experience. Developed by Schubert et al., this questionnaire was subsequently translated into Chinese and validated for reliability and validity by Liang Jiahui et al. The results demonstrated its strong reliability and validity, with a Cronbach's α coefficient of 0.82. The Chinese version comprises 13 items organized into three dimensions: spatial presence (Items 2, 3, 9), involvement (Items 1, 6, 10), and realism (Items 4, 5, 8, 11, 12, 13). Item 7 reflects overall presence. Each item employs a 7-point Likert scale ranging from -3 to 3 points, with items 10 and 12 reverse-scored. The total score ranges from -39 to 39 points, where a higher score indicates a better sense of presence experience in the virtual reality environment.
  Item 7 reflects overall presence. Each item uses a 7-point Likert scale ranging from -3 to 3 points, with items 10 and 12 reverse-scored. The total score rang

CONTACTS AND LOCATIONS:
Locations (1):
- Nursing school of Fujian Medical university, Fujian, Fuzhou, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol